CLINICAL TRIAL: NCT03622645
Title: Developing An Objective Measurement Method With The Leap Motion Sensor For Hand And Wrist's Range Of Motion: Validity And Reliability Study
Brief Title: An Objective Measurement Method With The Leap Motion Sensor For Hand And Wrist's Range Of Motion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Saime Nilay Arman, Principal Investigator, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10840098-604
Record Dates: First submitted 2018-07-24; First posted 2018-08-09 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Range of Motion
Keywords: Range of motion; Wrist; Hand; Finger; Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Range of motion in hand (Experimental): Assessment of Wrist flexion/extension, radial/ulnar deviation, supination/pronation, 1.-5. DIP, PIP and MCP flexion/extension ROM measurements of the fingers with universal goniometer and Leap motion sensor
  Interventions: Device: Assessment of Range of Motion with Leap Motion sensor

INTERVENTIONS:
Device: Assessment of Range of Motion with Leap Motion sensor — An ROM measurement method called as HandROM by us will be developed with leap motion sensor

SUMMARY:
The aim of the study was to develop a low cost, clinically easy to use measurement method with the Leap motion sensor for objectively evaluating range of motion (ROM), and to investigate the validity and reliability of this application.

DETAILED DESCRIPTION:
. Wrist flexion / extension, radial / ulnar deviation, supination / pronation, 1.-5. of the fingers DIP, PIP and MCP flexion / extension ROM measurements will be made with universal goniometer and developed Leap motion sensor (LMC) based measurement method.

The study consists of two basic steps:

1. Development of measurement method with LMC Identification of normROM measurement procedure Identification of ROM measurement reporting Establishing the precursor version of the software of the measurement method Checking ROM measurement performance criteria and providing feedback Measuring the movement defined on 5 persons and providing feedback Creation of the last available version of the measurement method
2. Validity and reliability study Measurements of hand and wrist ROM with developed measurement method with LMC and universal goniometer for three times and calculation mean of three measurement for two methods

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* Have any hand/wrist problems between the ages of 18-40 years.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Range of Motion | Baseline
  Wrist flexion / extension, radial / ulnar deviation, supination / pronation, 1. -5. DIP, PIP and MCP flexion / extension EHA measurements of the fingers will be made with universal goniometer and developed Leap motion sensor based measurement method.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arman N, Oktay AB, Tarakci D, Tarakci E, Akgul YS. The validity of an objective measurement method using the Leap Motion Controller for fingers wrist, and forearm ranges of motion. Hand Surg Rehabil. 2021 Sep;40(4):394-399. doi: 10.1016/j.hansur.2021.03.007. Epub 2021 Mar 26. PMID 33781957